CLINICAL TRIAL: NCT02589509
Title: Cognitive Rehabilitation and Brain Activity of Attention-Control Impairment in TBI
Brief Title: Cognitive Rehabilitation and Brain Activity of Attention Control in TBI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No one was recruited
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N1920-P; I21RX001920-01A1 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-28 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Brain Injuries, Traumatic
Keywords: Event-related potentials; Attention; Cognitive rehabilitation; Independent activities of daily living
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct-Metacognitive (Experimental): Direct attention training followed by metacognitive strategy training
  Interventions: Behavioral: Direct-attention training using web-based BrainHQ; Behavioral: Goal Management Training (GMT)
- Metacognitive-Direct (Experimental): Metacognitive strategy training followed by direct-attention training
  Interventions: Behavioral: Direct-attention training using web-based BrainHQ; Behavioral: Goal Management Training (GMT)

INTERVENTIONS:
Behavioral: Direct-attention training using web-based BrainHQ — BrainHQ (by Posit Science Corp.) computerized attention training using the following modules: "Divided attention," "Target tracker," "Double Decision," "Mixed Signals," and "Freeze Frame."
Behavioral: Goal Management Training (GMT) — A compensatory metacognitive strategy-based intervention program that teaches strategies for improving attentional control and problem solving.

SUMMARY:
The purpose of this study is to test an innovative combination of direct-attention training and metacognitive training in the treatment of attention impairments in Veterans with moderate-to-severe traumatic brain injury (TBI) who report experiencing attentional problems. Enrolled participants will be randomized to receive either the direct-attention training or metacognitive training first and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods of 4 weeks and a post-treatment 4 weeks later. In addition to the rehabilitation treatments, participants will also perform measures of complex functional activities (e.g., independent activities of daily living or IADLs) and neurocognitive tests of attention-control functions. Participants will also perform an attentional task that probes the function of three different attentional systems while brain wave activity (i.e., electroencephalography or EEG) is being recorded in order to assess changes in brain function that may be improved by the rehabilitation approach. Planned enrollment will be 36 Veterans.

DETAILED DESCRIPTION:
Attention impairment is ubiquitous in TBI survivors. This is a devastating impairment because attention is the backbone of cognitive systems. Attention is requisite for other cognitive processes that are vital to everyday functioning such as memory, problem solving, language skills, and the cognitive control of behavior. Studies of attention training have shown improved attention on laboratory measures, but limited translation to real-world tasks. Notably, these previously-tested rehabilitation approaches have not included training in the very cognitive processes needed for translation of training to everyday tasks which include internal verbalization and self-monitoring, also called metacognitive strategies. One training method for metacognitive strategies has shown promise, but is lacking in basic attention training. Rehabilitation specialists have recently argued for a rehabilitation approach wherein both basic foundational attention and metacognitive strategies should be synergistically combined. Consequently, the investigators will test an innovative combination of direct-attention training and metacognitive training for which the other compensates disadvantages of each. Because of the promise of each type of training separately, and the potential additive effects of the combination, it is critical to test this combined attention and metacognitive training in Veteran survivors of chronic moderate-to-severe traumatic brain injury (TBI). The investigators will address the following two specific aims: the investigators propose to conduct a pilot study to examine cognitive rehabilitation therapy (CRT) effects in a group of Veterans with chronic moderate to severe TBI (m/sTBI), focused on remediating attention-control impairments using both direct-attention and metacognitive-strategy training approaches in a AB/BA crossover design with 1-month follow-up to address the following two specific aims: 1) Test treatment response to combined direct-attention and metacognitive-strategy training in Veterans with chronic m/sTBI; and 2) identify mechanisms and biomarkers of rehabilitation-related neuroplasticity. Under the first aim the investigators will test for effects of combined direct-attention and metacognitive-strategy training on measures of complex functional activities and neurocognitive tests of attention-control functions. Under the second aim, the investigators will test effects of the their CRT approach on behavioral and brain activity while participants perform a well-validated attentional task that probes the function of three dissociable attentional systems. The approach is innovative because it combines a theoretically motivated and novel approach to address a significant source of disability in Veteran survivors of TBI. The proposed research is significant because findings will form the foundation for a larger-scale trial to enable us to determine the durability of gains and the functional impact of treatment on Veteran's real world activities and to more positively shape healthcare for our Veterans who are suffering from TBI. Outcome measures will include standardized tests of neurocognitive functioning such as attention and other cognitive skills, measures of self care, ability to live independently, social role participation, life satisfaction, TBI-related quality of life, mood/anxiety, and attention-related scalp-recorded brain event-related potentials (ERPs, derived from electroencephalography).

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF/OND Veterans with moderate or severe TBI as described by DOD/VA common definition.
* Self-report of attentional problems, confirmed with psychometric testing.
* Ruff 2 & 7 selective attention task score <= 1.5 standard deviations from demographically-matched norms.
* Able to participate in study at 12-60 months post injury without contraindications.
* Age 21-55 years.
* Willingness to be randomized and to participate in treatment procedures.
* Capacity to visit the laboratory for repeated treatment and testing sessions.
* Access to internet-enabled home computer.
* English as Native language.
* Adequate reading comprehension to allow completion of study-related questionnaires.
* Reliable digit span (RDS) score > 7.

Exclusion Criteria:

* Pre-existing neurological disorder associated with cerebral dysfunction (e.g., stroke, history of epilepsy or chronic seizure disorder).
* Current alcohol or drug use/dependence.
* Pre-existing severe psychiatric disorder (e.g., schizophrenia, bipolar disorder) or history of psychiatric diagnosis sufficiently severe to have resulted in inpatient hospitalization.
* Current suicidal or homicidal ideation.
* Reported involvement in current litigation.
* Reported history of pre-injury learning disability.
* Not competent to provide written informed consent (i.e., not able to demonstrate understanding or expectations of study and potential risks of participation).
* Does not fully understand the nature of the study and requirements of participation.
* Does not understand task instructions.
* Validity testing score on RDS <= 7.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Timed Instrumental Activities of Daily Living (TIADL) | Baseline TIADL Reaction Time assessed pretreatment
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) | Change from Baseline in TIADL Reaction Time assessed at 8 weeks
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) | Change from Baseline in TIADL Reaction Time assessed at 12 weeks (1-month post treatment)
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) - Accuracy | Change from Baseline in TIADL Accuracy assessed at 4 weeks
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) - Accuracy | Change from Baseline in TIADL Accuracy assessed at 8 weeks
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) - Accuracy | Change from Baseline in TIADL Accuracy assessed at 12 weeks (1 month post treatment)
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Ability Score | Change from Baseline in MPAI-4 Ability Score assessed at 4 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Ability Score | Change from Baseline in MPAI-4 Ability Score assessed at 8 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Ability Score | Change from Baseline in MPAI-4 Ability Score assessed at 12 weeks (1 month post treatment)
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Adjustment Score | Change from Baseline in MPAI-4 Adjustment Score assessed at 4 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Adjustment Score | Change from Baseline in MPAI-4 Adjustment Score assessed at 8 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Adjustment Score | Change from Baseline in MPAI-4 Adjustment Score assessed at 12 weeks (1 month post treatment)
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Participation Score | Change from Baseline in MPAI-4 Participation Score assessed at 4 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Participation Score | Change from Baseline in MPAI-4 Participation Score assessed at 8 weeks
  Assesses global outcome, including ability, adjustment and community participation indices.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Participation Score | Change from Baseline in MPAI-4 Participation Score assessed at 12 weeks (1 month post treatment)
  Assesses global outcome, including ability, adjustment and community participation indices.
Timed Instrumental Activities of Daily Living (TIADL) - Reaction Time score | Baseline (pretreatment) on TIADL - Reaction Time score
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Timed Instrumental Activities of Daily Living (TIADL) - Accuracy score | Baseline (pretreatment) on TIADL - Accuracy score
  The TIADL is a timed, performance-based measure of everyday cognition/instrumental activities of daily living (IADLs) in which participants are presented with common everyday stimuli (e.g., medication labels, transportation schedules, cake-mix ingredients, phone book) and asked to answer questions. The dependent variables are the number of accurate responses and response speed to each accurate item is recorded.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) | Baseline (pretreatment) MPAI-4 Adjustment score
  Assesses global outcome, including ability, adjustment and community participation indices. The MPAI-4 is a 35-item questionnaire-based inventory that will be completed study staff and TBI survivors. It offers three subscales (Ability, Adjustment, and Participation) and has well-documented psychometric properties. MPAI-4 items represent the range of physical, cognitive, emotional, behavioral, and societal problems that TBI survivors often encounter; it also assess major obstacles to community integration.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) | Baseline (pretreatment) MPAI-4 Participation score
  Assesses global outcome, including ability, adjustment and community participation indices. The MPAI-4 is a 35-item questionnaire-based inventory that will be completed study staff and TBI survivors. It offers three subscales (Ability, Adjustment, and Participation) and has well-documented psychometric properties. MPAI-4 items represent the range of physical, cognitive, emotional, behavioral, and societal problems that TBI survivors often encounter; it also assess major obstacles to community integration.
Attention Network Test (ANT) Alerting Reaction Time score | Change from Baseline in Altering Reaction Time Score assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Alerting Reaction Time score | Change from Baseline in Altering Reaction Time Score assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Alerting Reaction Time score | Change from Baseline in Altering Reaction Time Score assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Orient Reaction Time score | Baseline (pretreatment) Orienting Reaction Time score
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Orienting Reaction Time score | Change from Baseline in Orienting Reaction Time Score assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Orienting Reaction Time score | Change from Baseline in Orienting Reaction Time Score assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Orienting Reaction Time score | Change from Baseline in Orienting Reaction Time Score assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Executive-Control Reaction Time score | Baseline (pretreatment) Executive-Control Reaction Time score
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Executive-Control Reaction Time score | Change from Baseline in Executive-Control Reaction Time Score assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Executive-Control Reaction Time score | Change from Baseline in Executive-Control Reaction Time Score assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Executive-Control Reaction Time score | Change from Baseline in Executive-Control Reaction Time Score assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Attention Network Test (ANT) Alerting Reaction Time score | Baseline (pretreatment) Alerting Reaction Time score
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Alerting Amplitude | Baseline ANT ERP (N1) Alerting Amplitude assessed pretreatment
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Alerting Amplitude | Change from Baseline in ANT ERP (N1) Alerting Amplitude assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Alerting Amplitude | Change from Baseline in ANT ERP (N1) Alerting Amplitude assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Alerting Amplitude | Change from Baseline in ANT ERP (N1) Alerting Amplitude assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Orienting Amplitude | Baseline ANT ERP (N1) Orienting Amplitude assessed pretreatment
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Orienting Amplitude | Change from Baseline in ANT ERP (N1) Orienting Amplitude assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Orienting Amplitude | Change from Baseline in ANT ERP (N1) Orienting Amplitude assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (N1) Orienting Amplitude | Change from Baseline in ANT ERP (N1) Orienting Amplitude assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (P3) Executive Amplitude | Baseline ANT ERP (P3) Executive Amplitude assessed pretreatment
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (P3) Executive Amplitude | Baseline ANT ERP (P3) Executive Amplitude assessed at 4 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (P3) Executive Amplitude | Baseline ANT ERP (P3) Executive Amplitude assessed at 8 weeks
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
ANT ERP (P3) Executive Amplitude | Baseline ANT ERP (P3) Executive Amplitude assessed at 12 weeks (1 month post treatment)
  The ANT combines a covert cueing paradigm with a classic flanker task to behaviorally probe independent but interactive components of attention in a single experimental paradigm. Scalp-recorded electroencephalography (EEG) will be acquired from 64 sensors while participants perform the ANT to derive event-related potentials (ERPs) reflecting alerting, orienting, and executive-control components of attention and enable probing of brain plasticity associated with attention rehabilitation.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Ability Score | Baseline MPAI-4 Ability Score assessed pretreatment
  Assesses global outcome, including ability, adjustment and community participation indices. The MPAI-4 is a 35-item questionnaire-based inventory that will be completed study staff and TBI survivors. It offers three subscales (Ability, Adjustment, and Participation) and has well-documented psychometric properties. MPAI-4 items represent the range of physical, cognitive, emotional, behavioral, and societal problems that TBI survivors often encounter; it also assess major obstacles to community integration.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Adjustment Score | Baseline MPAI-4 Adjustment Score assessed pretreatment
  Assesses global outcome, including ability, adjustment and community participation indices. The MPAI-4 is a 35-item questionnaire-based inventory that will be completed study staff and TBI survivors. It offers three subscales (Ability, Adjustment, and Participation) and has well-documented psychometric properties. MPAI-4 items represent the range of physical, cognitive, emotional, behavioral, and societal problems that TBI survivors often encounter; it also assess major obstacles to community integration.
Mayo-Portland Adaptability Inventory, 4th edition (MPAI-4) - Participation Score | Baseline MPAI-4 Participation Score assessed pretreatment
  Assesses global outcome, including ability, adjustment and community participation indices. The MPAI-4 is a 35-item questionnaire-based inventory that will be completed study staff and TBI survivors. It offers three subscales (Ability, Adjustment, and Participation) and has well-documented psychometric properties. MPAI-4 items represent the range of physical, cognitive, emotional, behavioral, and societal problems that TBI survivors often encounter; it also assess major obstacles to community integration.

SECONDARY OUTCOMES:
Mindful Attention Awareness Scale-Lapses Only (MAAS-LO) | Change from Baseline in MAAS-LO Score assessed at 4 weeks
  The MAAS-LO is a 12-item 6-point Likert-type scale designed to measure everyday attentional lapses (infrequent to very frequent).
Mindful Attention Awareness Scale-Lapses Only (MAAS-LO) | Change from Baseline in MAAS-LO Score assessed at 8 weeks
  The MAAS-LO is a 12-item 6-point Likert-type scale designed to measure everyday attentional lapses (infrequent to very frequent).
Mindful Attention Awareness Scale-Lapses Only (MAAS-LO) | Change from Baseline in MAAS-LO Score assessed at 12 weeks (1 month post treatment)
  The MAAS-LO is a 12-item 6-point Likert-type scale designed to measure everyday attentional lapses (infrequent to very frequent).
Satisfaction with Life Scale (SWLS) | Baseline SWLS Score assessed pretreatment
  The SWLS assesses patient's perceived satisfaction with life. It is a 5-item 7-point Likert-type scale with a range from "strongly disagree" to "strongly agree." The total score is used as a measure of satisfaction with life.
Mindful Attention Awareness Scale-Lapses Only (MAAS-LO) | Baseline (pretreatment) on MAAS-LO
  The MAAS-LO is a 12-item 6-point Likert-type scale designed to measure everyday attentional lapses (infrequent to very frequent).
Satisfaction with Life Scale (SWLS) | Change from Baseline in SWLS Score assessed at 4 weeks
  The SWLS assesses patient's perceived satisfaction with life. It is a 5-item 7-point Likert-type scale with a range from "strongly disagree" to "strongly agree." The total score is used as a measure of satisfaction with life.
Satisfaction with Life Scale (SWLS) | Change from Baseline in SWLS Score assessed at 8 weeks
  The SWLS assesses patient's perceived satisfaction with life. It is a 5-item 7-point Likert-type scale with a range from "strongly disagree" to "strongly agree." The total score is used as a measure of satisfaction with life.
Satisfaction with Life Scale (SWLS) | Change from Baseline in SWLS Score assessed at 12 weeks (1 month post treatment)
  The SWLS assesses patient's perceived satisfaction with life. It is a 5-item 7-point Likert-type scale with a range from "strongly disagree" to "strongly agree." The total score is used as a measure of satisfaction with life.

OTHER OUTCOMES:
Ruff 2 & 7 Selective Attention Task (RSAT) | Eligibility screening (Pretreatment)
  Psychometric validation/measurement of participant's subjective complaint of attention disturbance
Reliable Digit Span (RDS) | Eligibility screening (Pretreatment)
  The Reliable Digit Span (RDS) test, scored from the forward and backward digit span from the Wechsler Adult Intelligence Scale version 4 (WAIS-IV), will be used to determine the potential presence of suboptimal effort; cutoff for the RDS will be a score 7.
Mental Health Screening Form 3rd edition (MHSF-III) | Eligibility screening (Pretreatment)
  The MHSF-III is a structured interview that will be used to screen for the presence of exclusionary major psychopathology.
Wide Range Achievement Test, 4th edition (WRAT-4; word-reading subtest) | Group matching (Pretreatment)
  The word-reading subtest of the WRAT-4 will administered to obtain a measure of estimated premorbid cognitive functioning, and groups will be matched, on average, for scores on this test.

CONTACTS AND LOCATIONS:
Overall Officials: William M Perlstein, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No